CLINICAL TRIAL: NCT04819854
Title: A First-in Man, Phase I Study Investigating the Safety and Tolerability of EP395 in Healthy Volunteers
Brief Title: Single and Multiple Ascending Dose Study With EP395
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpiEndo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EP395-001
Record Dates: First submitted 2021-03-04; First posted 2021-03-29 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Adult ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Single and multiple ascending doses
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded, placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EP395 (Experimental): EP395 in ascending doses. Orally, once daily.
  Interventions: Drug: EP395
- Placebo (Placebo Comparator): Placebo, weight matched in ascending doses. Orally, once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EP395 — capsule for oral treatment
  Arms: EP395
Drug: Placebo — capsule for oral treatment
  Arms: Placebo

SUMMARY:
This is a study to asses the safety and tolerability of single and multiple ascending doses of EP395, administered by oral capsules, in healthy subjects with the aim to determine the safe dose range of EP395 for further clinical development

DETAILED DESCRIPTION:
This is a study to asses the safety and tolerability of single and multiple ascending doses of EP395, administered by oral capsules, in healthy subjects with the aim to determine the safe dose range of EP395 for further clinical development. The study consists of two parts, part A where single-ascending doses will be assessed and part B where multiple-ascending doses will be assessed. The primary objective being safety and tolerability as well as the pharmacokinetic properties of EP395.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedures.
2. Able to understand and comply with the requirements of the study, as judged by the investigator or designee.
3. Men and women between 18-65 years inclusive
4. Female subjects must either be of non-childbearing potential or if of childbearing potential, must not be pregnant or breast feeding and use a highly effective birth control method during treatment and for 90 days following last dose
5. Male subjects must use highly effective contraception during treatment and for 90 days following last administered dose
6. Subject must agree not to donate semen or ova/oocytes during the study and for 90 days after the last dose of IMP
7. Body mass index (BMI) ≥ 18 and ≤ 32 kg/m2.
8. Subjects with normal hearing
9. Subjects must be in good health at the time of screening

Exclusion Criteria:

1. History or presence of any clinically relevant acute or chronic medical or psychiatric condition that could interfere with the subject's safety.
2. History or presence of vestibular disorder including vertigo, dizziness or other auditory impairment as judged by the investigator or designee.
3. After 10 minutes supine rest at the time of screening or prior to dosing, any vital signs values outside the following ranges:

   * Systolic blood pressure <90 or >150 mmHg, or
   * Diastolic blood pressure <50 or >95 mmHg, or
   * Pulse <40 or >90 bpm
4. Any clinically significant abnormalities in resting ECG at the time of screening or pre-dose Day 1 including prolonged QTcF (>450 ms for males; >470 ms for females) and cardiac arrhythmias, as judged by the Investigator or designee.
5. Clinically significant abnormalities in renal function:

   * serum creatinine >ULN
   * eGFR <60 mL/min or ≥ 60mL/min with evidence of any kidney dysfunction (e.g. proteinuria, or clinical findings as judged by the investigator)
6. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP (Day 1).
7. Malignancy within the past five years with the exception of in situ removal of basal cell carcinoma or resected benign colonic polyps.
8. Any planned major surgery within the duration of the study.
9. History of latent or active tuberculosis or a positive Quantiferon test at screening.
10. Females who are pregnant, breast feeding or plan to be pregnant during the study period or 90 days after.
11. Female subjects with a positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at screening and within 24 h prior to the first administration of IMP.
12. Positive serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus (HIV) 1 and/or 2 antibodies at screening.
13. Positive PCR test for active COVID -19 tested within seven days prior to administration of the IMP on Day 1.
14. History of any drug and/or alcohol abuse in the past two years prior to screening.
15. Regular alcohol consumption in males >21 units per week and females >14 units per week.
16. Positive urine drugs of abuse test and/or alcohol breath test at screening or on admission to the unit prior to administration of the IMP on Day -1 that cannot be accounted for by concomitant medication in the opinion of the Investigator or designee.
17. Current or previous use of tobacco, nicotine products or e-cigarettes in the past six months.
18. Smoking history of > 5 pack years.
19. Positive urine cotinine test at screening or Day -1.
20. Use of any prescribed or non-prescribed medication including analgesics, herbal remedies, vitamins and minerals within two weeks prior to the (first) administration of IMP, except those listed below, at the discretion of the Investigator or designee:

    * hormone replacement therapy (HRT)
    * hormonal contraception
    * occasional intake of paracetamol (maximum 2000 mg/day for 3 consecutive days)
    * nasal decongestants without cortisone for a maximum of 10 days
    * antihistamines for a maximum of 10 days
    * anticholinergics for a maximum of 10 days
21. Use of antacids, PPIs or any medication that changes gastric pH within two weeks prior to the first administration of IMP (Day 1).
22. Use of macrolide antibiotics within two weeks prior to the first administration of IMP (Day 1)
23. Subjects who have received a live vaccine in the 28 days prior to Day 1.
24. Plasma donation within one month of screening or blood donation (or corresponding blood loss) ≥400mL during the three months prior to screening.
25. Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator or designee at screen.
26. Subject has dietary restrictions incompatible with the diet that can be provided by the study site, in the opinion of the Investigator or is unwilling to refrain from consuming restricted foods and beverages during the study
27. Regular excessive caffeine consumption defined by a daily intake of >5 cups of caffeine containing beverages.
28. Known history of intolerance or hypersensitivity to macrolides, EP395 or to any other component of the formulation.
29. Known history of intolerance to lactose.
30. Clinically significant serious adverse reaction, allergy or serious hypersensitivity, including to any drug or food, as judged by the Investigator or designee.
31. Involvement in the planning and conduct of the study (applies to all EpiEndo, CRO or investigational site staff).
32. Participation in another clinical study with an experimental drug within three months or 5 half-lives, whichever is shorter, before the administration of IMP.
33. Considered unsuitable for entry into the study in any other way at the discretion of the principal investigator or designee, e.g. investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
To assess the safety of EP395 | from baseline to day 7 and day 42
  Adverse Events
To assess the effect of EP395 on ECG | from baseline to day 7 and day 42
  QT intervals
To assess the effect of EP395 on temperature | from baseline to day 7 and day 42
  Temperature
To assess the effect of EP395 on blood pressure | from baseline to day 7 and day 42
  Blood pressure
To assess the effect of EP395 on pulse | from baseline to day 7 and day 42
  Pulse
To assess the effect of EP395 on hearing | from baseline to day 7 and day 42
  Audiometry

SECONDARY OUTCOMES:
To assess the Cmax of EP395 in plasma and blood | from baseline to day 7 and day 42
  Maximum Plasma Concentration [Cmax]
To assess the tmax of EP395 in plasma and blood | from baseline to day 7 and day 42
  Time to reach Cmax (Tmax)
To assess the t½ of EP395 in plasma and blood | from baseline to day 7 and day 42
  Time to half-life (t½)
To assess the AUC of EP395 in plasma and blood | from baseline to day 7 and day 42
  Area Under the Curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, Prof., Principal Investigator — The Medicines Evaluation Unit (MEU) Ltd.
Locations (1):
- The Medicines Evaluation Unit (MEU) Ltd., Manchester, United Kingdom